CLINICAL TRIAL: NCT01084005
Title: A Phase III Randomised, Double Blind, Placebo-controlled, Parallel Group, Efficacy and Safety Study of Linagliptin (5 mg) Administered Orally Once Daily Over 24 Weeks in Type 2 Diabetic Patients (Age >= 70 Years) With Insufficient Glycaemic Control( HbA1c >= 7.0) Despite Metformin and/or Sulphonylurea and/or Insulin Therapy
Brief Title: Efficacy and Safety of Linagliptin in Elderly Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.63; 2009-015255-25 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- linagliptin (Experimental): patients receive linagliptin 5 mg tablets once daily
  Interventions: Drug: linagliptin
- placebo (Placebo Comparator): patients receive placebo tablets matching linagliptin 5 mg once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: linagliptin — patients receive linagliptin 5 mg tablets once daily
  Arms: linagliptin
Drug: placebo — patients receive placebo matching linagliptin 5 mg once daily
  Arms: placebo

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of linagliptin (5 mg / once daily) compared to placebo given for 24 weeks as add-on therapy to stable treatment in elderly patients with T2DM with insufficient glycaemic control

ELIGIBILITY:
Inclusion criteria:

1. Type 2 diabetes mellitus
2. HbA1c >= 7.0%
3. Age >= 70 years
4. Signed and dated written informed consent

Exclusion criteria:

1. Myocardial infarction, stroke or TIA within 3 months prior to informed consent
2. Impaired hepatic function
3. Treatment with glitazones, GLP-1 analogues, DPP-4 inhibitors or rapid acting or pre-mixed insulins
4. Treatment with anti-obesity drugs

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (34):
- Australia (7):
  - 1218.63.61005 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 1218.63.61006 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 1218.63.61003 Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - 1218.63.61002 Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - 1218.63.61007 Boehringer Ingelheim Investigational Site, East Ringwood, Victoria
  - 1218.63.61001 Boehringer Ingelheim Investigational Site, Parkville, Victoria
  - 1218.63.61004 Boehringer Ingelheim Investigational Site, Reservoir, Victoria
- Canada (8):
  - 1218.63.10008 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.63.10003 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.63.10005 Boehringer Ingelheim Investigational Site, Hawkesbury, Ontario
  - 1218.63.10007 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1218.63.10006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.63.10001 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1218.63.10002 Boehringer Ingelheim Investigational Site, Saint Romuald, Quebec
  - 1218.63.10004 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Denmark (8):
  - 1218.63.45007 Boehringer Ingelheim Investigational Site, Aalborg
  - 1218.63.45002 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1218.63.45003 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1218.63.45001 Boehringer Ingelheim Investigational Site, Birkerød
  - 1218.63.45008 Boehringer Ingelheim Investigational Site, Hellerup
  - 1218.63.45006 Boehringer Ingelheim Investigational Site, Hillerød
  - 1218.63.45004 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1218.63.45005 Bispebjerg Hospital, København NV
- Netherlands (6):
  - 1218.63.31008 Boehringer Ingelheim Investigational Site, Beek en Donk
  - 1218.63.31007 Boehringer Ingelheim Investigational Site, Beerzerveld
  - 1218.63.31012 Boehringer Ingelheim Investigational Site, Doetinchem
  - 1218.63.31014 Boehringer Ingelheim Investigational Site, Etten-Leur
  - 1218.63.31009 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1218.63.31001 Boehringer Ingelheim Investigational Site, Tubbergen
- Sweden (5):
  - 1218.63.46004 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1218.63.46003 Boehringer Ingelheim Investigational Site, Järfälla
  - 1218.63.46001 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.63.46002 Boehringer Ingelheim Investigational Site, Sundsvall
  - 1218.63.46005 Boehringer Ingelheim Investigational Site, Uppsala

REFERENCES:
- [Derived] Lajara R, Aguilar R, Hehnke U, Woerle HJ, von Eynatten M. Efficacy and safety of linagliptin in subjects with long-standing type 2 diabetes mellitus (>10 years): evidence from pooled data of randomized, double-blind, placebo-controlled, phase III trials. Clin Ther. 2014 Nov 1;36(11):1595-605. doi: 10.1016/j.clinthera.2014.07.020. Epub 2014 Sep 16. PMID 25236917
- [Derived] McGill JB, Barnett AH, Lewin AJ, Patel S, Neubacher D, von Eynatten M, Woerle HJ. Linagliptin added to sulphonylurea in uncontrolled type 2 diabetes patients with moderate-to-severe renal impairment. Diab Vasc Dis Res. 2014 Jan;11(1):34-40. doi: 10.1177/1479164113507068. Epub 2013 Oct 29. PMID 24169807
- [Derived] Barnett AH, Huisman H, Jones R, von Eynatten M, Patel S, Woerle HJ. Linagliptin for patients aged 70 years or older with type 2 diabetes inadequately controlled with common antidiabetes treatments: a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Oct 26;382(9902):1413-23. doi: 10.1016/S0140-6736(13)61500-7. Epub 2013 Aug 13. PMID 23948125
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/1218/1218.63_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 241 patients were randomised in a 2:1 ratio to receive treatment with linagliptin 5mg (n=162) or placebo (n=79). All randomised patients were treated.
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Linagliptin 5 mg: Patients randomized to receive treatment with Linagliptin 5mg
Period: Overall Study
Arm/Group | Placebo | Linagliptin 5 mg
Started | 79 | 162
Completed | 74 | 146
Not Completed | 5 | 16
Not completed — Adverse Event | 1 | 8
Not completed — Protocol Violation | 3 | 7
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 5 mg | Total
Number analyzed (Participants) | 79 | 162 | 241
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.9 (4.2) | 74.9 (4.4) | 74.9 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 46 | 76
  Male | 49 | 116 | 165
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 29.80 (4.54) | 29.60 (4.74) | 29.67 (4.67)
Glycosylated Hemoglobin A1 (HbA1c) [Mean (Standard Deviation); unit: Percent] — Based upon the full analysis set (FAS) with 78 and 160 patients
  Percent | 7.70 (0.70) | 7.82 (0.78) | 7.78 (0.76)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Based upon the FAS with 78 and 160 patients
  mg/dL | 144.1 (29.6) | 152.7 (28.7) | 149.9 (29.2)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline to Week 24
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and prior use of insulin.
Time Frame: Baseline and week 24
Population: FAS consisting of all randomised patients who were treated with at least one dose of study drug, had a baseline, and at least 1 on-treatment HbA1c measurement. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 160
Percent | 0.04 (0.07) | -0.61 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.64, 95% CI [-0.81 to -0.48], Standard Error of Mean 0.08

2. Secondary Outcome: HbA1c Change From Baseline to Week 6
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 6 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and prior use of insulin.
Time Frame: Baseline and week 6
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 160
Percent | -0.07 (0.05) | -0.42 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.35, 95% CI [-0.45 to -0.24], Standard Error of Mean 0.05

3. Secondary Outcome: HbA1c Change From Baseline to Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and prior use of insulin.
Time Frame: Baseline and week 12
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 160
Percent | -0.03 (0.06) | -0.60 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI [-0.71 to -0.43], Standard Error of Mean 0.07

4. Secondary Outcome: HbA1c Change From Baseline to Week 18
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and prior use of insulin.
Time Frame: Baseline and week 18
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 160
Percent | 0.04 (0.07) | -0.58 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.62, 95% CI [-0.77 to -0.47], Standard Error of Mean 0.08

5. Secondary Outcome: FPG Change From Baseline to Week 24
Description: This change from baseline reflects the Week 24 FPG minus the baseline FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and prior use of insulin.
Time Frame: Baseline and week 24
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 156
mg/dL | 10.1 (4.3) | -10.6 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -20.7, 95% CI [-30.2 to -11.2], Standard Error of Mean 4.8

6. Secondary Outcome: FPG Change From Baseline to Week 6
Description: This change from baseline reflects the Week 6 FPG minus the baseline FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and prior use of insulin, week repeated within patient and week by treatment interaction.
Time Frame: Baseline and week 6
Population: FAS Observed cases (OC)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 77 | 153
mg/dL | 4.6 (2.7) | -14.1 (2.0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -18.6, 95% CI [-24.7 to -12.6], Standard Error of Mean 3.1

7. Secondary Outcome: FPG Change From Baseline to Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and prior use of insulin, week repeated within patient and week by treatment interaction.
Time Frame: Baseline and week 12
Population: FAS (OC)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 75 | 148
mg/dL | 6.8 (2.9) | -14.7 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -21.5, 95% CI [-28.1 to -14.8], Standard Error of Mean 3.4

8. Secondary Outcome: FPG Change From Baseline to Week 18
Description: This change from baseline reflects the Week 18 FPG minus the baseline FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and prior use of insulin, week repeated within patient and week by treatment interaction.
Time Frame: Baseline and week 18
Population: FAS (OC)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 68 | 145
mg/dL | 9.6 (3.6) | -12.0 (2.5)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -21.6, 95% CI [-29.8 to -13.4], Standard Error of Mean 4.2

9. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 7%. Only patients with baseline HbA1c >= 7%
Time Frame: Baseline and week 24
Population: FAS with baseline HbA1c >=7% and non-completers considered as failure imputation (NCF)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 72 | 149
percentage of patients | 8.3 | 38.9
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 8.319, 95% CI [3.321 to 20.837]

10. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7% at week 24 were calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 7%.
Time Frame: Baseline and week 24
Population: FAS (NCF)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 160
percentage of patients | 11.5 | 41.9

11. Secondary Outcome: Percentage of Patients Who Have a HbA1c Lowering by at Least 0.5% at Week 24
Description: The percentage of patients with an HbA1c reduction of ≥0.5% at week 24 from baseline was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c reduction less than 0.5%
Time Frame: Baseline and week 24
Population: FAS (NCF)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 160
percentage of patients | 12.8 | 54.4

12. Secondary Outcome: Number of Patients With Rescue Therapy
Description: The use of rescue therapy was planned for patients failing to achieve preset criteria based on glucose levels during the randomised treatment period of the trial
Time Frame: week 24
Population: FAS (OC)
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 78 | 160
Number of patients | 11 | 7
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Lina 5 mg qd vs Placebo; Test type: Superiority or Other; p = 0.0048, Regression, Logistic; Odds Ratio (OR) = 0.214, 95% CI 2-sided [0.073 to 0.625]

ADVERSE EVENTS:
Time Frame: 24 weeks + 7 days of follow-up
Arm/Group | Placebo | Linagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 5/79 | 14/162
Other Adverse Events (participants affected / at risk) | 37/79 | 70/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Linagliptin 5 mg (N=162)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Vestibular neuronitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Linagliptin 5 mg (N=162)
Diarrhoea (Gastrointestinal disorders) | 2 | 9
Nasopharyngitis (Infections and infestations) | 7 | 17
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Urinary tract infection (Infections and infestations) | 5 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 13 | 37
Dizziness (Nervous system disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.